CLINICAL TRIAL: NCT04154761
Title: Resection of the Inferior Vena Cava Due to Tumor Involvement Allows Long-Term Survival in Different Neoplasms
Brief Title: Resection of the Inferior Vena Cava Due to Tumor Involvement
Acronym: CAVARESECT
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Infanta Cristina (Other)
Responsible Party: Principal Investigator, Diego López Guerra, Hepatobiliary Surgeon, Principal Investigator, Hospital Universitario Infanta Cristina
Other Study IDs: UE-CHUB 002-2019
Record Dates: First submitted 2019-11-05; First posted 2019-11-06 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Neoplasms; Surgery--Complications; Vascular Diseases; Vein Disease
Keywords: Inferior vena cava; radical resection; Vascular reconstruction
MeSH Terms: conditions — Neoplasms; Vascular Diseases | interventions — Plastic Surgery Procedures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Resection of inferior vena cava and reconstruction — Resection of inferior vena cava and reconstruction with primary repair, resection with autologous or prosthetic patch repair, and circumferential resection with graft replacement

SUMMARY:
The involvement of the inferior vena cava (IVC) in advanced abdominal tumors is a surgical challenge, given the high postoperative morbidity and poor long-term prognosis. The goal was to analyze the experience, perioperative management, and results.

Investigators have evaluated short and long-term results of surgical resections of tumors with associated inferior vena cava resection performed between 2012 and 2018.

DETAILED DESCRIPTION:
Data Collection:

Investigators retrospectively looked at patients who, from January 2012 to December 2018, underwent surgical procedures in the unit for IVC-specific tumors or for IVC resections due to secondary infiltrative tumors. In some cases, the IVC involvement was an intraoperative finding.

Patients with primary or secondary IVC involvement who underwent surgery were included in the study. Patients with metastasis found during intraoperative exploration were excluded from the study.

Diagnostic management included establishment of a medical history, performance of clinical examination and imaging tests, including an abdominal ultrasound and computerized tomography (CT) scan, to confirm the tumor origin and growth, as well as infiltration, if any, of adjacent structures. These also allowed to rule out distant metastases, and to assess resectability and the option for vascular reconstruction. In some cases, the decision to resect the IVC was made during surgery, because IVC involvement was an intraoperative finding which remained unknown up to that point.

The variables taken into account were age, sex, BMI, the American Society of Anesthesiologists (ASA) classification, tumor type, preoperative chemotherapy and/or radiation therapy. In addition, another variable considered was whether the finding was intraoperative or preoperative. Perioperative clinical results, surgical approach, type of IVC resection and reconstruction, and intraoperative complications were recorded. Details of the postoperative course were collected. Some of the key short-term data recorded included length of hospital stay, complications' ranking (according to the Clavien-Dindo score; 'severe complication' is defined as greater or equal to IIIa), re-operation, re-admission and operative mortality (< 90 days after operation). Some of the key long-term data recorded were patency of IVC or prosthesis (as determined by a CT scan), neoadjuvant and adjuvant chemotherapy, specific disease-free survival and overall survival (OS).

Surgical Approach Management of IVC involvement was categorized in three groups, according to the surgical repair necessary: resection with primary repair, resection with autologous or prosthetic patch repair, and circumferential resection with graft replacement. Primary repair was defined as resection of a portion of the IVC with primary closure when <50% narrowing of the lumen would result. Patch closure was planned when a larger defect created by the resection required patch repair to avoid narrowing of the IVC. Circumferential resection of the IVC was managed with replacement using a prosthetic graft.

For surgical planning, investigators used the classification according to Kulayat, which subdivides the IVC into three segments: upper portion (level 1)-extending from the opening of the hepatic veins up to the right atrium-, middle portion (level 2)-extending from the renal veins to the hepatic veins-, and lower portion (level 3)-extending from the junction of the iliac veins to the opening of the renal veins.

Intravenous heparin was not used during the clamping time of the IVC. Heparinized saline (2units/ml of heparin sodium) was used, however, to flush out the prosthesis if being used for reconstruction. A therapeutic heparin dose is used for 30 days after surgery, and patients with prosthesis receive oral blood thinners for at least six months.

Follow-up Patient follow-up included measuring tumor markers and performing a chest-abdominal CT scan every three months for the first two years; then, twice a year; and then, annually, after five years. Local recurrence was defined as a return of a tumor within the surgical field, whereas systemic recurrence was defined as recurrent disease outside said field.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary or secondary IVC involvement who underwent surgery.

Exclusion Criteria:

* Patients with metastasis found during intraoperative exploration.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who, from January 2012 to December 2018, underwent surgical procedures in our unit for IVC-specific tumors or for IVC resections due to secondary infiltrative tumors.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Complication | 90 days
  Surgical complications rates
Overall survival | 5 years
  Patients overall survival after resection

CONTACTS AND LOCATIONS:
Locations (1):
- Diego López-Guerra, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: Undecided